CLINICAL TRIAL: NCT05978310
Title: The Effect of Patient Position on Cerebral Regional Oxygen Saturation in Intracranial Surgeries
Brief Title: NIRS and Anesthesiology
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Trakya University (Other)
Responsible Party: Principal Investigator, Ars Gor Dr Oguzhan Gulgen, Research assistant doctor, Trakya University
Other Study IDs: Trakya U/Anesthesiology
Record Dates: First submitted 2023-07-28; First posted 2023-08-07 (Actual); Last update posted 2023-08-07 (Actual); Status verified 2023-07

CONDITIONS: NIRS and Anesthesiology

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Group P: Patients operated in the prone position
- Group S: Patients operated in the supine position
- Group L: Patients operated in the lateral position

SUMMARY:
Our aim in this study is to investigate the effects of the positions applied in Intracranial Surgery on Cerebral Oxygenation(with NIRS device) and to evaluate the superiority of the patient positions used to each other.

DETAILED DESCRIPTION:
One of the main goals during anesthesia practice is to provide adequate tissue oxygenation. For this purpose, many parameters such as ECG, blood pressure, blood gas, and urine monitoring are monitored. However, it is a serious deficiency that the brain, which is the most sensitive organ to ischemia, is not monitored in intracranial surgeries . Trying to keep the intraoperative blood gas parameters and cerebral blood flow at normal values in order to overcome this deficiency brings along serious problems in proportion to the frequency of the measurement interval. For this reason, evaluation of tissue oxygenation with the Near Infrared Spectroscopy (NIRS) method has come to the fore in recent years, and especially cerebral regional oxygen saturation (rSo2) follow-ups have begun to be performed more frequently. The values obtained by this method represent 75% venous, 20% arterial and 5% capillary compartment of the measurement area .

While deciding on the positions applied in intracranial surgery, it may be necessary to apply modifications by keeping the surgical application site in the foreground. The preferred patient position in the operation can help prevent complications and serious side effects. Although each position applied in intracranial operations has advantages and disadvantages, the surgeon should choose the most suitable position for the patient and pathology. The "park bench" position is widely used in posterior fossa operations and has replaced the sitting position for most neurosurgical procedures . However, since the advantages of the sitting position could not be obtained, this position was also changed and the modified Park bench position with 30 degrees upside tilt was used. This position can provide similar advantages with the sitting position and also reduces the risk of venous air embolism and hypotension . The modified sitting position for posterior fossa surgery versus the semi-sitting or "beach chair" position retains many of the advantages and provides a rapid trendelenburg in case of air embolism. The classical sitting position causes postural hypotension in approximately 1/3 of the patients and severe hypotension is seen in 2-5% of the patients. Excellent surgical intervention, drier area and less blood loss, reduced facial swelling are the advantages of the sitting position. However, the risk of venous air embolism and increased pneumocephalus should not be ignored.

In addition to the hemodynamic changes due to all these known positions, there is no follow-up of cerebral regional oxygen saturation (rSo2) monitoring depending on the position, which we could not detect in the literature. This monitoring can contribute to the optimal continuation of cerebral blood flow while deciding on the appropriate position of the patients. In this case, the postoperative mortality and morbidity of the patients can be reduced. In addition, intraoperative cerebral oxygenation monitoring is critical for predicting delirium in the postoperative period.

Our aim in this study is to investigate the effects of the positions applied in Intracranial Surgery on Cerebral Oxygenation and to evaluate the superiority of the patient positions used to each other.

ELIGIBILITY:
Inclusion Criteria:

* Patients who will undergo intracranial surgery
* Patients aged 25-75 years
* Patients in the ASA I-II-III risk group

Exclusion Criteria:

* Patients with a GCS below 15
* patients with heart failure, renal failure, liver failure
* patients with congenital neurological deficits
* patients who cannot be contacted

Ages: 25 Years to 75 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: 150 patients in the ASA I-II-III risk group between the ages of 25-75 who will undergo intracranial surgery at Trakya University Medical Faculty Hospital will be included in the study.
Sampling Method: Probability Sample
Enrollment: 150 (Estimated)
Dates: Start 2022-10-01 (Actual); Primary Completion 2025-01-01 (Estimated); Study Completion 2025-02-01 (Estimated)

PRIMARY OUTCOMES:
NIRS values | October 1, 2022 /February 1, 2025

CONTACTS AND LOCATIONS:
Locations (1):
- Trakya university, Edirne, Turkey (Türkiye)